CLINICAL TRIAL: NCT05849311
Title: A Randomized, Double-blind, Single-dose, Parallel Controlled Phase I Study to Evaluate the Pharmacokinetics, Safety, and Immunogenicity of Envafolimab in Healthy Male Subjects Before and After the Manufacturing Process Change
Brief Title: Phase I Trial of Envafolimab for Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: 3D Medicines (Sichuan) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: 3D Medicines (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: KN035-CN-BE
Record Dates: First submitted 2023-04-27; First posted 2023-05-08 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2023-07

CONDITIONS: Healthy Male
MeSH Terms: interventions — envafolimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Envafolimab with new manufacturing process (Experimental): 80 healthy male subjects with Envafolimab with new manufacturing process
  Interventions: Drug: Envafolimab with new manufacturing process
- Envafolimab with old manufacturing process (Active Comparator): 80 healthy male subjects with Envafolimab with old manufacturing process
  Interventions: Drug: Envafolimab with old manufacturing process

INTERVENTIONS:
Drug: Envafolimab with new manufacturing process — Dosage form:
  Envafolimab is a monoclonal antibody drug administered subcutaneously in a minimum packaging unit of 1.0 ml solution in a single-use glass vial containing a total of 200 mg of Envafolimab.
  Treatment method:
  Envafolimab, single dose, 1 mg/kg, subcutaneously.
  Arms: Envafolimab with new manufacturing process
Drug: Envafolimab with old manufacturing process — Dosage form:
  Envafolimab is a monoclonal antibody drug administered subcutaneously in a minimum packaging unit of 1.0 ml solution in a single-use glass vial containing a total of 200 mg of Envafolimab.
  Treatment method:
  Envafolimab, single dose, 1 mg/kg, subcutaneously.
  Arms: Envafolimab with old manufacturing process

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic similarity, safety, and immunogenicity of Envafolimab in healthy male subjects before and after the manufacturing process change.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to fully read, understand, and sign the informed consent form;
2. Male subjects aged 18-45 years
3. Clinical examinations in the screening period are normal or abnormal without clinical significance;
4. A body mass index (BMI) in the range of 19 to 26 kg/m22, and a body weight between 50 and 85 kg;
5. Use effective contraceptive methods from the beginning of the informed consent to 5 months after the use of the drug, and have no plans to give birth or donate sperm.

Exclusion Criteria:

1. Systolic blood pressure ≥140 mmHg/ diastolic blood pressure ≥90 mmHg or systolic blood pressure < 90 mmHg/ diastolic blood pressure < 60 mmHg, pulse > 100 beats /min or < 50 beats /min at screening or baseline examination;
2. QT interval (QTcF) ≥450;
3. Estimated glomerular filtration rate eGFR < 90 ml/min/1.73m2;
4. Thyroid function beyond the normal range;
5. ALT > ULN Or AST > ULN;
6. Prior treatment with a PD-1/L1 inhibitor;
7. Have taken any prescription drug, over-the-counter drug, any vitamin product or herbal or health product within 14 days prior to study drug administration;
8. Had a history of upper respiratory tract infection or other acute infection within 14 days prior to study drug administration;
9. Positive hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus antibody or syphilis.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
AUC0-t | From pre-dose to day 85
  Area under the plasma concentration-time curve
Cmax | From pre-dose to day 85
  concentration

SECONDARY OUTCOMES:
AUC0-infinity | From pre-dose to day 85
  Area under the plasma concentration-time curve
Tmax | From pre-dose to day 85
  Time to maximum concentration
CL | From pre-dose to day 85
  Clearance
λz | From pre-dose to day 85
  Apparent terminal elimination rate constant
t1/2 | From pre-dose to day 85
  Half-life (
Vd | From pre-dose to day 85
  Volume of distribution
Safety and tolerance | From pre-dose to day 85
  Adverse events (AE)
Immunogenicity assessment | From pre-dose to day 85
  Anti-drug Antibody (ADA)

CONTACTS AND LOCATIONS:
Overall Officials: Qing He, Principal Investigator — Beijing Goboard Boren Hospital
Locations (1):
- Beijing Gaobo Boren Hosipital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided